CLINICAL TRIAL: NCT02342314
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3143753 and LY3185643 in Healthy Subjects
Brief Title: A Study of LY3143753 and LY3185643 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15503; I7U-MC-GAHA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY3143753 (Part A) (Experimental): Single subcutaneous (SC) injection of ascending doses of LY3143753 on Day 1
  Interventions: Drug: LY3143753 (Part A)
- LY3185643 (Part B) (Experimental): Single SC injection of ascending doses of LY3185643 on Day 1
  Interventions: Drug: LY3185643 (Part B)
- Placebo (Part A) (Placebo Comparator): Single SC injection of normal saline on Day 1
  Interventions: Drug: Placebo (Part A and Part B)
- rGlucagon (Part B) (Active Comparator): Single SC injection on Day 1
  Interventions: Drug: rGlucagon (Part B)
- Placebo (Part B) (Placebo Comparator): Single SC injection of normal saline on Day 1
  Interventions: Drug: Placebo (Part A and Part B)

INTERVENTIONS:
Drug: LY3143753 (Part A) — Administered via SC injection
  Arms: LY3143753 (Part A)
Drug: LY3185643 (Part B) — Administered via SC injection
  Arms: LY3185643 (Part B)
Drug: Placebo (Part A and Part B) — Administered via SC injection
  Arms: Placebo (Part A); Placebo (Part B)
Drug: rGlucagon (Part B) — Administered via SC injection
  Arms: rGlucagon (Part B)

SUMMARY:
The study involves a single dose of LY3143753 or LY3185643, given as an injection into the abdomen. The study will evaluate the effects of the LY3143753 or LY3185643 on your body. The study is approximately 12 weeks for each participant, not including screening. Screening is required within 28 days prior to the start of the study. This study involves Part A (LY3143753) and Part B (LY3185643). Participants may only enroll in one part and at one dose level.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Are investigator site personnel directly affiliated with this study and their immediate families
* Are currently enrolled in a clinical trial involving an investigational product (IP) or off-label use of a drug or device
* Have participated, within the last 3 months, in a clinical trial
* Have known or ongoing psychiatric disorders
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* History of/current phaeochromocytoma
* History of/current insulinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Part A): Single subcutaneous (SC) injection of normal saline on Day 1.
- 0.05 mg of LY3143753 (Part A): Part A: 0.05 milligram (mg) of LY3143753 given as a single SC injection on Day 1.
- 0.1 mg of LY3143753 (Part A): Part A: 0.1 mg of LY3143753 given as a single SC injection on Day 1.
- 0.2 mg of LY3143753 (Part A): Part A: 0.2 mg of LY3143753 given as a single SC injection on Day 1.
- 0.4 mg of LY3143753 (Part A): Part A: 0.4 mg of LY3143753 given as a single SC injection on Day 1.
- 1.0 mg of LY3143753 (Part A): Part A: 1.0 mg of LY3143753 given as a SC injection on Day 1.
- Placebo (Part B): Part B: Single SC injection of normal saline on Day 1.
- 0.01 mg of LY3185643 (Part B): Part B: 0.01 mg of LY3185643 given as a single SC injection on Day 1.
- 0.03 mg of LY3185643 (Part B): Part B: 0.03 mg of LY3185643 given as a single SC injection on Day 1.
- 0.05 mg of LY3185643 (Part B): Part B: 0.05 mg of LY3185643 given as a single SC injection on Day 1.
- 0.06 mg of LY3185643 (Part B): Part B: 0.06 mg of LY3185643 given as a single SC injection on Day 1.
- 0.1 mg of LY3185643 (Part B): Part B: 0.1 mg of LY3185643 given as a single SC injection on Day 1.
- 0.2 mg of LY3185643 (Part B): Part B: 0.2 mg of LY3185643 given as a single SC injection on Day 1.
- 0.3 mg of LY3185643 (Part B): Part B: 0.3 mg of LY3185643 given as a single SC injection on Day 1.
- 0.48 mg of LY3185643 (Part B): Part B: 0.48 mg of LY3185643 given as a single SC injection on Day 1.
- 0.72 mg of LY3185643 (Part B): Part B: 0.72 mg of LY3185643 given as a single SC injection on Day 1.
- rGlucagon (Part B): Part B: 1.0 mg of rGlucagon given as a single SC injection. (Part B).
Period: Part A
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A) | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B) | rGlucagon (Part B)
Started | 6 | 3 | 3 | 3 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 3 | 3 | 3 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A) | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B) | rGlucagon (Part B)
Started | 0 (Participants received placebo in Part A.) | 0 (Participants received LY3143753 in Part A.) | 0 (Participants received LY3143753 in Part A.) | 0 (Participants received LY3143753 in Part A.) | 0 (Participants received LY3143753 in Part A.) | 0 (Participants received LY3143753 in Part A.) | 11 (Participants received placebo in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 3 (Participants received LY3185643 in Part B.) | 6 (Participants received rGlucagon in Part B.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY3143753 (Part A) | LY3185643 (Part B) | Total
Number analyzed (Participants) | 24 | 44 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 17 | 40 | 57
  >=65 years | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 17 | 37 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 44 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 23 | 41 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 24 | 44 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Baseline to Study Completion (Up to 84 Days)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Part A); Placebo (Part B): Single SC injection on Day 1.
- 0.05 mg of LY3143753 (Part A): 0.05 mg of LY3143753 given as a single SC injection.
- 0.1 mg of LY3143753 (Part A): 0.1 mg of LY3143753 given as a single SC injection.
- 0.2 mg of LY3143753 (Part A): 0.2 mg of LY3143753 given as a single SC injection.
- 0.4 mg of LY3143753 (Part A): 0.4 mg of LY3143753 given as a single SC injection.
- 1 mg of LY3143753 (Part A): 1 mg of LY3143753 given as a single SC injection.
- 0.01 mg of LY3185643 (Part B): 0.01 mg of LY3185643 given as a single SC injection on Day 1.
- 0.03 mg of LY3185643 (Part B): 0.03 mg of LY3185643 given as a single SC injection on Day 1.
- 0.05 mg of LY3185643 (Part B): 0.05 mg of LY3185643 given as a single SC injection on Day 1.
- 0.06 mg of LY3185643 (Part B): 0.06 mg of LY3185643 given as a single SC injection on Day 1.
- 0.1 mg of LY3185643 (Part B): 0.1 mg of LY3185643 given as a single SC injection on Day 1.
- 0.2 mg of LY3185643 (Part B): 0.2 mg of LY3185643 given as a single SC injection on Day 1.
- 0.3 mg of LY3185643 (Part B): 0.3 mg of LY3185643 given as a single SC injection on Day 1.
- Part B 0.48 mg of LY3185643: 0.48 mg of LY3185643 given as a single SC injection on Day 1.
- 0.72 mg of LY3185643 (Part B): 0.72 mg of LY3185643 given as a single SC injection on Day 1.
- r Glucagon (Part B): 1 mg of rGlucagon given as a single SC injection. (Part B).
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1 mg of LY3143753 (Part A) | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | Part B 0.48 mg of LY3185643 | 0.72 mg of LY3185643 (Part B) | r Glucagon (Part B)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 6 | 3 | 11 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of Part A
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4, 6, 8 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- 0.05 mg of LY3143753 (Part A): 0.05 mg of LY3143753 given as a single SC injection on Day 1.
- 0.1 mg of LY3143753 (Part A): 0.1 mg of LY3143753 given as a single SC injection on Day 1.
- 0.2 mg of LY3143753 (Part A): 0.2 mg of LY3143753 given as a single SC injection on Day 1.
- 0.4 mg of LY3143753 (Part A): 0.4 mg of LY3143753 given as a single SC injection on Day 1.
- 1.0 mg of LY3143753 (Part A): 1.0 mg of LY3143753 given as a single SC injection on Day 1.
Arm/Group | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3
nanogram/milliliter (ng/mL) | 0.726 (81) | 1.05 (73) | 2.95 (13) | 5.73 (47) | 11.4 (38)

3. Secondary Outcome: PK: Cmax of Part B
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4, 6, 8 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 0.48 mg of LY3185643 (Part B): 0.48 mg of LY3185643 given as a single SC injection on Day 1.
Arm/Group | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
ng/mL | 0.126 (12) | 0.367 (51) | 1.19 (70) | 0.951 (32) | 2.34 (48) | 4.25 (53) | 4.67 (51) | 6.49 (58) | 9.67 (14)

4. Secondary Outcome: PK: Area Under the Concentration Curve From Zero to Infinity (AUC[0-∞]) of Part A
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4, 6, 8 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3
nanogram*hour/milliliter (ng*hr/mL) | 1.44 (46) | 1.57 (97) | 5.76 (38) | 12.6 (33) | 22.6 (62)

5. Secondary Outcome: PK: AUC(0-∞) of Part B
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4, 6, 8 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
ng*hr/mL | NA (NA) — PK data from 3 participants at this lowest LY3185643 dose was very limited with few measurable data points which led to the inability to estimate the AUC(0-infinity) PK parameter. | 0.564 (8) | 2.61 (42) | 1.34 (24) | 3.73 (22) | 8.87 (18) | 10.8 (14) | 16.2 (55) | 21.5 (9)

6. Secondary Outcome: PK: Time to Maximum Drug Concentration (Tmax) of Part A
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4, 6, 8 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3
hour | 0.67 [0.67 to 1.00] | 0.83 [0.33 to 1.00] | 0.67 [0.67 to 0.67] | 1.04 [0.67 to 1.50] | 1.25 [0.67 to 1.25]

7. Secondary Outcome: PK: Tmax of Part B
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4, 6, 8 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
hour | 0.83 [0.83 to 0.83] | 0.67 [0.50 to 1.00] | 0.83 [0.83 to 1.00] | 0.67 [0.55 to 0.83] | 0.50 [0.50 to 1.00] | 1.25 [1.00 to 1.25] | 1.23 [0.83 to 1.25] | 1.75 [0.67 to 1.75] | 0.83 [0.67 to 1.00]

8. Secondary Outcome: Pharmacodynamic (PD): Absolute Maximum Blood Glucose of Part A
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4 Hours
Population: All participants who received at least one dose of study drug or placebo and have evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram/deciliter (mg/dL)
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 6 | 3
milligram/deciliter (mg/dL) | 101 (10) | 168 (26) | 197 (17) | 179 (13) | 188 (10) | 177 (19)

9. Secondary Outcome: PD Absolute Maximum Blood Glucose of Part B
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4 Hours
Population: All participants who received at least one dose of study drug or placebo and have evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Groups:
- Part B 0.72 mg of LY3185643 (Part B): 0.72 mg of LY3185643 given as a single SC injection on Day 1.
- 1.0 mg of rGlucagon (Part B): 1.0 mg of rGlucagon given as a single SC injection.
Arm/Group | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | Part B 0.72 mg of LY3185643 (Part B) | 1.0 mg of rGlucagon (Part B)
Number analyzed (Participants) | 11 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
mg/dL | 95.1 (5) | 103 (11) | 98.1 (10) | 128 (36) | 117 (7) | 167 (16) | 186 (7) | 146 (16) | 192 (16) | 188 (3) | 162 (11)

10. Secondary Outcome: PD: Maximum Glucose Increase (Gmax) of Part A
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A)
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 6 | 3
mg/dL | 4.14 (112) | 66.1 (63) | 103 (17) | 84.9 (18) | 91.5 (20) | 79.8 (40)

11. Secondary Outcome: PD: Gmax of Part B
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Groups:
- 1.0 mg of rGlucagon (Part B): 1.0 mg of rGlucagon given as a single SC injection. (Part B).
Arm/Group | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B) | 1.0 mg of rGlucagon (Part B)
Number analyzed (Participants) | 10 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
mg/dL | 4.69 (54) | 7.2 (12.6) | 5.04 (189) | 28.1 (144) | 21.8 (66) | 76.1 (35) | 89.4 (14) | 58.4 (35) | 102 (25) | 105 (6) | 71.8 (23)

12. Secondary Outcome: PD: Time to Maximum Blood Glucose (Gtmax) of Part A
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data.
Measure: Median (Full Range); unit: hour
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 6 | 3
hour | 0.96 [0.00 to 4.00] | 1.00 [0.75 to 1.00] | 1.00 [0.58 to 1.00] | 0.67 [0.5 to 0.67] | 0.79 [0.75 to 2.5] | 0.58 [0.50 to 1.33]

13. Secondary Outcome: PD: Gtmax of Part B
Time Frame: Predose, 5,10, 15, 20, 25, 30, 35, 40, 45, 50, 550, 60, 70, 80, 90, 105, minutes and 2, 2.5, 3, 4 Hours
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data.
Measure: Median (Full Range); unit: hour
Arm/Group | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B) | 1.0 mg of rGlucagon (Part B)
Number analyzed (Participants) | 11 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
hour | 0.5 [0.0 to 1.5] | 0.5 [0.0 to 0.5] | 0.67 [0.25 to 0.83] | 1.0 [0.83 to 1.33] | 0.67 [0.67 to 0.75] | 0.75 [0.75 to 1.17] | 1.17 [0.92 to 1.33] | 0.58 [0.5 to 0.75] | 1.17 [0.83 to 1.33] | 0.75 [0.67 to 1.0] | 0.46 [0.33 to 0.75]

14. Secondary Outcome: QT Interval as Corrected by the Fridericia Method (QTcF) Change From Baseline of Part A
Time Frame: Baseline, 8 hours after drug administration
Population: All randomized participants who received at least one dose of study drug and who had evaluable QTcF data.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Groups:
- 0.1 mg of LY3143753 (Part A): 0.01 mg of LY3143753 given as a single SC injection on Day 1.
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1.0 mg of LY3143753 (Part A)
Number analyzed (Participants) | 6 | 2 | 3 | 2 | 5 | 3
milliseconds (msec) | 0.6 (6.4) | NA (NA) — Data was not available for one participant at each of these time points so the mean and standard deviation (SD) were not applicable. | 0.2 (18.6) | NA (NA) — Data was not available for one participant at each of these time points so the mean and SD were not applicable. | 6.1 (14.5) | 6.1 (13.3)

15. Secondary Outcome: QTcF Change From Baseline of Part B
Time Frame: Baseline, 8 hours after drug administration
Population: All randomized participants who received at least one dose of study drug and had evaluable QTcF data.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Groups:
- rGlucagon (Part B): 1 mg of rGlucagon given as a single SC injection. (Part B).
Arm/Group | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | 0.48 mg of LY3185643 (Part B) | 0.72 mg of LY3185643 (Part B) | rGlucagon (Part B)
Number analyzed (Participants) | 9 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 6
milliseconds (msec) | -1.4 (8.3) | -2.9 (8.5) | -10.2 (3.3) | -5.9 (12.5) | -4.1 (7.8) | 0.5 (11.3) | -4.7 (7.6) | 2.5 (13.0) | -2.1 (2.7) | NA (NA) — Data was not available for one participant at each of these time points so the mean and SD were not applicable. | -7.7 (5.8)

ADVERSE EVENTS:
Arm/Group | Placebo (Part A) | 0.05 mg of LY3143753 (Part A) | 0.1 mg of LY3143753 (Part A) | 0.2 mg of LY3143753 (Part A) | 0.4 mg of LY3143753 (Part A) | 1 mg of LY3143753 (Part A) | Placebo (Part B) | 0.01 mg of LY3185643 (Part B) | 0.03 mg of LY3185643 (Part B) | 0.05 mg of LY3185643 (Part B) | 0.06 mg of LY3185643 (Part B) | 0.1 mg of LY3185643 (Part B) | 0.2 mg of LY3185643 (Part B) | 0.3 mg of LY3185643 (Part B) | Part B 0.48 mg of LY3185643 | 0.72 mg of LY3185643 (Part B) | r Glucagon (Part B)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/3 | 1/6 | 1/3 | 1/11 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 2/3 | 3/3 | 3/3 | 4/6 | 3/3 | 5/11 | 3/3 | 1/3 | 1/3 | 2/3 | 3/3 | 3/3 | 2/3 | 3/3 | 3/3 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=6) | 0.05 mg of LY3143753 (Part A) (N=3) | 0.1 mg of LY3143753 (Part A) (N=3) | 0.2 mg of LY3143753 (Part A) (N=3) | 0.4 mg of LY3143753 (Part A) (N=6) | 1 mg of LY3143753 (Part A) (N=3) | Placebo (Part B) (N=11) | 0.01 mg of LY3185643 (Part B) (N=3) | 0.03 mg of LY3185643 (Part B) (N=3) | 0.05 mg of LY3185643 (Part B) (N=3) | 0.06 mg of LY3185643 (Part B) (N=3) | 0.1 mg of LY3185643 (Part B) (N=3) | 0.2 mg of LY3185643 (Part B) (N=3) | 0.3 mg of LY3185643 (Part B) (N=3) | Part B 0.48 mg of LY3185643 (N=3) | 0.72 mg of LY3185643 (Part B) (N=3) | r Glucagon (Part B) (N=6)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=6) | 0.05 mg of LY3143753 (Part A) (N=3) | 0.1 mg of LY3143753 (Part A) (N=3) | 0.2 mg of LY3143753 (Part A) (N=3) | 0.4 mg of LY3143753 (Part A) (N=6) | 1 mg of LY3143753 (Part A) (N=3) | Placebo (Part B) (N=11) | 0.01 mg of LY3185643 (Part B) (N=3) | 0.03 mg of LY3185643 (Part B) (N=3) | 0.05 mg of LY3185643 (Part B) (N=3) | 0.06 mg of LY3185643 (Part B) (N=3) | 0.1 mg of LY3185643 (Part B) (N=3) | 0.2 mg of LY3185643 (Part B) (N=3) | 0.3 mg of LY3185643 (Part B) (N=3) | Part B 0.48 mg of LY3185643 (N=3) | 0.72 mg of LY3185643 (Part B) (N=3) | r Glucagon (Part B) (N=6)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days